CLINICAL TRIAL: NCT05611424
Title: An Open-label, Single-center, Dose-escalation Clinical Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of FT-003 in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: Gene Therapy for Wet AMD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Frontera Therapeutics (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other); Tianjin Medical University Eye Hospital (Other); Peking Union Medical College Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT003WA-1
Record Dates: First submitted 2022-11-02; First posted 2022-11-10 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Neovascular Age-related Macular Degeneration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- FT003 Dose 1 (Experimental): Low dose of FT-003
  Interventions: Genetic: FT-003
- FT003 Dose 2 (Experimental): Mid dose of FT-003
  Interventions: Genetic: FT-003
- FT003 Dose 3 (Experimental): High dose of FT-003
  Interventions: Genetic: FT-003

INTERVENTIONS:
Genetic: FT-003 — Administered via intraocular injection.

SUMMARY:
FT-003 is a gene therapy product developed for the treatment of neovascular age-related macular degeneration (nAMD). Neovascular AMD is the main cause of blindness among elderly individuals. The available therapies for treating nAMD require life-long intravitreal (IVT) injections every 4-12 weeks to maintain efficacy. Administration of FT-003 has the potential to treat nAMD by providing durable expression of therapeutic levels of intraocular protein and maintaining the vision of patients. FT-003 is designed to reduce the current treatment burden which often results in undertreatment and vision loss in patients with nAMD receiving anti-VEGF therapy in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that are willing and able to follow study procedures;
* Female or male patients ≥45 years old at the time of signing the ICF;
* Clinically diagnosed with nAMD;
* Presence of active CNV
* The best corrected visual acuity (BCVA) of the studied eye is ≤ 53 letters;

Exclusion Criteria:

• Presence of any other intraocular diseases other than nAMD in the studied eye that would affect the improvement of visual acuity and require treatment during the study for prevention or treatment of visual loss, as judged by the investigator.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability after FT-003 injection | At Week 52
  Incidence and severity of AE (Common Terminology Criteria for Adverse Events 5.0)

SECONDARY OUTCOMES:
Changes in best-corrected visual acuity (BCVA) of the studied eye from baseline | At Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Peirong Lu, Professor, Principal Investigator — The First Affiliated Hospital of Soochou University; Xiaorong Li, Professor, Principal Investigator — Tianjin Medical University Eye Hospital; Hanyi Min, Principal Investigator — Peking Union Medical College Hospital; Guangming Wan, Principal Investigator — The First Affiliated Hospital of Zhengzhou University

IPD SHARING:
Plan to Share IPD: No